CLINICAL TRIAL: NCT01023399
Title: A Nested Open Labeled Study to Compare the Effectiveness and Safety of a Fixed-dose Combination of Artesunate Plus Amodiaquine (ASAQ Winthrop®) in the Unsupervised Treatment of Uncomplicated Plasmodium Falciparum Malaria Attacks in Two Patient Groups Enrolled at Two Year-intervals in a Pilot District of Côte d'Ivoire
Brief Title: Artesunate Plus Amodiaquine in Malaria in Cote d'Ivoire
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Medicines for Malaria Venture (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARAMF_L_04314
Record Dates: First submitted 2009-12-01; First posted 2009-12-02 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2015-02

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria | interventions — amodiaquine, artesunate drug combination

ARMS (1):
- Artesunate + Amodiaquine (Experimental): Oral fixed combination of artesunate (AS) and amodiaquine (AQ)
  Once daily, dose according to age
  Infants 2-11 months: AS 25/AQ 67,5 mg (3 tablets/ blister)
  Toddlers 1-5 years: AS 50/AQ 135 mg (3 tablets/ blister)
  Children: 6-13 years: AS 100/AQ 270 mg (3 tablets/ blister)
  Adults: >= 14 years: AS 100/AQ 270 mg (6 tablets/ blister)
  3 day-treatment
  Interventions: Drug: Artesunate + Amodiaquine

INTERVENTIONS:
Drug: Artesunate + Amodiaquine — Artesunate + Amodiaquine fixed dose combination

SUMMARY:
The primary objective of this study is to demonstrate the non-inferiority of Polymerase Chain Reaction (PCR)-adjusted adequate clinical and parasitological response to artesunate plus amodiaquine at Day 28 in two groups of patients treated at the beginning of an artesunate plus amodiaquine implementation program and 24 months later.

The secondary objectives are Clinical and biological tolerability Evolution of gametocyte carriage Proportion of patients without fever at Day 3 Proportion of patients without parasite at Day 3 Treatment compliance Impact of implementation on anemia Measure of parasite sensibility to amodiaquine

ELIGIBILITY:
Inclusion Criteria:

* Body weight >=5kg
* Plasmodium falciparum infection with parasite density > 2000/µL
* Fever or history of fever
* Able to be treated by oral route
* No signs of severe malaria
* No known allergy to study drugs
* No other severe illnesses or underlying diseases
* No known pregnancy or negative urinary pregnancy test for women of child bearing age
* No participation in another ongoing clinical study

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 580 (Actual)
Dates: Start 2009-11; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Polymerase chain reaction (PCR)-corrected and uncorrected clinical and parasitological cure rate (ACPR) | Day 28

SECONDARY OUTCOMES:
Number of patients without fever | Day 3
Number of patients without parasite | Day 3
Number of gametocytes | Day 3, Day 7, Day 14, Day 21 and Day 28
Evolution of in vitro resistance rate | Day 3, Day 7, Day 14, Day 21 and Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational Site Number 1, Agboville District, Côte d’Ivoire

REFERENCES:
- [Derived] Assi SB, Nguessan AF, Aba YT, Toure AO, Menan H, Yavo JC, San KM, Bissagnene E, Duparc S, Lameyre V, Tanoh MA. Sustained Effectiveness of a Fixed-Dose Combination of Artesunate and Amodiaquine in 480 Patients with Uncomplicated Plasmodium falciparum Malaria in Cote d'Ivoire. Malar Res Treat. 2017;2017:3958765. doi: 10.1155/2017/3958765. Epub 2017 Dec 7. PMID 29362685